CLINICAL TRIAL: NCT00929812
Title: The Mechanisms Underlying the Glucagon-Induced Suppression of Ghrelin Secretion
Brief Title: Glucagon Modulation of Ghrelin Secretion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Ayman M Arafat, Dr.med., Charite Campus Benjamin Franklin
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: GluGhr-study 01082005; EudoraCT 2005-003714-15; Prüfplancode 01082005; BfArM 61-3910-4031020; EK EA4/108/05
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Healthy Subjects; Obesity; Diabetes Mellitus, Type 1
Keywords: obesity; food intake; glucagon; ghrelin; glucose; insulin
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucagon hydrochloride (Active Comparator): GlucaGen® 1 mg/1 ml intramuscularly
  Interventions: Drug: Glucagon hydrochloride (GlucaGen®)
- Placebo (Placebo Comparator): 1 ml NaCl 0.9%
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Glucagon hydrochloride (GlucaGen®) — 1 mg/1 ml of glucagon hydrochloride intramuscularly
  Other Names: GlucaGen® (Novo Nordisk Pharma, MA:28288.00.00)
  Arms: Glucagon hydrochloride
Drug: NaCl 0.9% — 1 ml NaCl 0.9% intramuscularly
  Arms: Placebo

SUMMARY:
As a counterregulatory hormone for insulin, glucagon plays a critical role in maintaining glucose homeostasis in vivo. It is well known that intramuscular glucagon administration stimulates growth hormone (GH), adrenocorticotropic hormone (ACTH) and cortisol release in humans. Recently, it has been shown that glucagon induces a remarkable decrease in ghrelin levels. The mechanisms underlying this effect are unclear and the role of changes in glucose, insulin, glucagon-like peptide-1 (GLP-1) and catecholamines are widely discussed. The aim of the present study is to further evaluate the effect of glucagon on ghrelin secretion and the possible role of the above mentioned factors in mediating this effect.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18 and < 60 years old.
* Patients with diabetes type 1 should fulfill the following criteria:

  * ICT Insulin therapy was necessary within the first 3 months after diagnosis;
  * HbA1c-Wert < 7%.

Exclusion Criteria:

* Diabetes type 1 or 2 (for the healthy group).
* Biochemical evidence of impaired hepatic or renal function.
* History of cardiovascular disease.
* Uncontrolled hypertension.
* Current inflammatory, malignant or psychiatric disease.
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Changes in satiety scale, total and acylated ghrelin concentrations. | During 240 min after Glucagon/Placebo administration.

SECONDARY OUTCOMES:
Changes in glucose, insulin and NEFA concentrations. | During 240 min after Glucagon/Placebo administration.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman M Arafat, Dr.med., Principal Investigator — Charite Campus Benjamin Franklin
Locations (1):
- Charite Campus Benjamin Franklin, Berlin, Germany

REFERENCES:
- [Background] Arafat AM, Perschel FH, Otto B, Weickert MO, Rochlitz H, Schofl C, Spranger J, Mohlig M, Pfeiffer AF. Glucagon suppression of ghrelin secretion is exerted at hypothalamus-pituitary level. J Clin Endocrinol Metab. 2006 Sep;91(9):3528-33. doi: 10.1210/jc.2006-0225. Epub 2006 Jun 20. PMID 16787987
- [Derived] Arafat AM, Weickert MO, Adamidou A, Otto B, Perschel FH, Spranger J, Mohlig M, Pfeiffer AF. The impact of insulin-independent, glucagon-induced suppression of total ghrelin on satiety in obesity and type 1 diabetes mellitus. J Clin Endocrinol Metab. 2013 Oct;98(10):4133-42. doi: 10.1210/jc.2013-1635. Epub 2013 Aug 21. PMID 23966238